CLINICAL TRIAL: NCT00480688
Title: A Study of the Immunogenicity of M. Bovis BCG, Delivered Intradermally in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB001
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2007-05-31 (Estimated); Status verified 2007-05

CONDITIONS: TB
Keywords: TB; BCG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: BCG

SUMMARY:
To assess the immunogenicity of M. bovis BCG, given intrademally in the standard dose used in clinical practice and to measure the development of the immune response in the first six months after administration. M. bovis BCG is a fully licensed vaccine that has been in routine clinical use for the last 50 years. It is the most widely administered vaccine in the world today and has an excellent safety record.

DETAILED DESCRIPTION:
Volunteers for the study will be recruited through advertisements. Each volunteer will have received an information sheet concerning the study and will have agreed to participate in writing.

Volunteers will be given at least 48 hours between reading the information leaflet and agreeing to participate. Female volunteers will have a pregnancy test prior to enrollment. Volunteers will give signed consent for their GP's to be notified about their participation in the trial. The GP will be faxed a letter on the day of screening and asked to reply if they know of a reason why the volunteer should not take part. The signed consent form will also be faxed with the letter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-65 years.
* Normal medical history and physical examination.
* Normal urine dipstick, blood count, liver enzymes, and creatinine.

Exclusion Criteria:

* Exposure to TB/BCG vaccination at any point. Previous residence in a TB endemic area.
* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy,immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder,liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
* Oral or systemic steroid medication or the use of immunosuppressive agents.
* Positive HIV or core HBV antibody test.
* Positive Heaf test
* Positive ANA or serum anti-DNA antibody.
* Confirmed pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2001-11; Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Induction of T cell responses | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen I McShane, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, CCVTM, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Result] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839